CLINICAL TRIAL: NCT02043041
Title: Explaining the Differences in HIV Prevalence and Incidence Between Black and White Men Who Have Sex With Men in Atlanta
Brief Title: Evaluation of the Quality of Self-collected Blood Spot Specimens for Laboratory HIV Testing - An InvolveMENt Sub Study
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Patrick S Sullivan, Professor, Emory University
Other Study IDs: IRB00042405; P30AI050409 (NIH)
Record Dates: First submitted 2014-01-21; First posted 2014-01-23 (Estimated); Last update posted 2015-06-25 (Estimated); Status verified 2015-06

CONDITIONS: HIV

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Dried blood spots will be collected and inspected for quality. Once quality is determined, samples will be destroyed. No identifying information will be associated with the sample.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1 Dried Blood Spot (DBS): Number of DBS Spots Participants will be asked to fill one spot on a dried blood spot collection card.
  Interventions: Other: Number of DBS Spots
- 3 DBS Spots: Number of DBS Spots Participants will be asked to fill three spots on a dried blood spot collection card.
  Interventions: Other: Number of DBS Spots
- 5 DBS Sports: Number of DBS Spots Participants will be asked to fill five spots on a dried blood spot collection card.
  Interventions: Other: Number of DBS Spots

INTERVENTIONS:
Other: Number of DBS Spots — The number of DBS spots on the card constitutes the experimental condition.

SUMMARY:
We will invite a convenience sample of up to 45 enrolled subjects to participate in an optional, self-administered blood specimen collection procedure to determine optimal procedures for collection.

DETAILED DESCRIPTION:
Participants will be recruited to this one-time assessment during their follow-up visits. After completing a consent procedure specific to this study component, participants will be provided with instructions on how to fully self-administer the procedure of a finger stick and also blotting to collect a blood specimen using a 1, 3 or 5 blood spot specimen collection card. These specimens will be labeled with the participant's unique identification number, and no other identifying information. The dried blood spots will be evaluated by a laboratorian to assess quality, but will not be tested for HIV. This evaluation will help determine what number of self-collected dried blood spots yields the highest usable quantity of sample for HIV testing. There will be a separate monetary incentive of $30 for this procedure.

ELIGIBILITY:
Inclusion Criteria:

* Must be either currently enrolled or previously enrolled in the InvolveMENt Study through Emory University
* Over 18 years old
* HIV Negative

Exclusion Criteria:

* Not enrolled or previously enrolled in the InvolveMENt Study through Emory University
* Under 18 years old
* HIV Positive

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be enrolled or previously enrolled in the InvolveMENt Study through Emory University. They will be assesed for study interest either at the end of their scheduled appointment with InvolveMENt, or will be contacted if consent to contact them for future studies was previously obtained through InvolveMENt.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Viable sample for HIV Testing | Outcome measure will be assessed with in two weeks of all samples being collected
  Samples will be examined and not tested by a lab technician for acceptability for HIV testing.

CONTACTS AND LOCATIONS:
Overall Officials: AD McNaghten, PHD, MHSA, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States